CLINICAL TRIAL: NCT03077048
Title: Short-term Metabolic Effects of Ketosteril® Supplemented Low Protein Diet in Pre-dialysis CKD Patients - A Randomized, Controlled, Open-labelled Clinical Trial
Brief Title: Short-term Metabolic Effects of Ketosteril® Supplemented Low Protein Diet in Pre-dialysis Chronic Kidney Disease (CKD) Patients
Acronym: CKD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Collaborators: EastHORN Clinical Services in CEE (Unknown); MLM Medical Labs GmbH (Industry); ALS Czech Republic, s.r.o. (Unknown); PCG Clinical Services AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Keto-022-CP1; 2016-003854-34 (EudraCT Number)
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Renal Insufficiency, Chronic
Keywords: CKD; Ketosteril; keto-acids; ketoanalogues; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ketosteril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low protein diet (No Intervention): Low protein diet with 0.6 g protein/kg BW/day (20-30% high biological value) and an energy intake of 30-35 kcal/kg BW/day
- Supplemented low protein diet (Experimental): Ketosteril® supplemented low protein diet (sLPD), (1 tablet/5 kg BW/day) with 0.6 g protein/kg BW/day (20-30% high biological value) and an energy intake of 30-35 kcal/kg BW/day
  Interventions: Drug: Ketosteril®

INTERVENTIONS:
Drug: Ketosteril® — Patients will be randomised to receive isonitrogenous and isocaloric LPD providing 0.6 g protein/kg BW/day and an energy intake of 30-35 kcal/kg BW/day with (test group) or without (control group) intake of Ketosteril® (1 tablet/5 kg BW/day). The control group will get additional food protein to balance the nitrogen content of Ketosteril® The mainly vegetarian diet will be maintained for 10 days.
  Other Names: EV product code: PRD1170237
  Arms: Supplemented low protein diet

SUMMARY:
Supplementation of ketoanalogues of essential amino acids improves the protein quality of protein restricted diets without burdening the kidneys. The ketoanalogues are transaminated by aminotransferases to the corresponding amino acids by incorporating nitrogen from amino groups derived from endogenous amino acid degradation. Therefore, less nitrogen needs to be excreted and the kidney's workload is reduced.

The purpose of the trial is to investigate the impact of Ketosteril® supplementation on A) nutritional safety and tolerance of a low protein diet (LPD) (0.6 g protein/kg bodyweight (BW)/day)and B) net protein synthesis in pre-dialysis CKD patients.

Changes of urea in serum and urine will be assessed under controlled metabolic balance conditions in non-dialysed CKD patients consuming a LPD supplemented with Ketosteril® at 1 tablet/5 kg body weight/day compared to the same, isonitrogenous and isocaloric diet without Ketosteril®.

Changes in protein synthesis and degradation at the defined protein intake with or without Ketosteril® supplementation will be investigated - based on nitrogen balance, normalized protein catabolic rates as well as blood levels of defined proteins as surrogate markers for net protein synthesis and anabolic signaling.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Non-dialysed male and female CKD patients with expected start of dialysis ≥ 3 months
3. eGFR ≥5 to < 30 ml/min/1.73 m2
4. Stable renal function at least 12 weeks before enrollment, defined by change in serum creatinine ≤ 80 µmol/L
5. Body mass index (BMI): ≥ 22 kg/m² and ≤ 35 kg/m2
6. Age: ≥ 40 to ≤ 75 years
7. Eligible physical status of the patient for participation in the study upon assessment of the investigator based on medical history, physical examination and clinical laboratory parameters

Exclusion Criteria:

1. Existing gastrointestinal diseases or pathological findings (e.g. heart, liver, or lung failure), which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient (e.g. persistent or frequent episodes of anorexia, vomiting, or diarrhea)
2. Active cancer
3. Diabetes treated with standard pharmacotherapy
4. HbA1c ≥ 48 mmol/mol, and/or fasting blood glucose ≥ 126 mg/dl (≥ 7 mmol/L))
5. Evidence of chronic infection or chronic inflammation; evidence of acute infection or acute inflammation
6. C-reactive protein (CRP) > 20 mg/L determined at screening examination
7. Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparation
8. Severe allergies or multiple drug allergies if judged as relevant for the clinical trial by the investigator
9. Patients suffering from hypercalcaemia with a serum calcium ≥ 2.9 mmol/L performed on screening examination
10. Major disorder of amino acid metabolism, e.g. hereditary diseases
11. Hospitalization within the previous 1 month
12. Proteinuria > 3 g/day
13. Regular intensive exercise
14. Ingestion of creatine supplements within the previous 1 month
15. Intake of other anabolic or anti catabolic agents within the previous 1 month
16. Any change of the chronic medication within 1 month before screening
17. Autosomal dominant polycystic kidney disease (ADPKD)
18. Positive anti-HIV-test (if positive to be verified by western blot), Hepatitis B surface antigen (HBsAG)-test (if positive to be verified by test for hepatitis B core antigen (HBc)- Immunoglobulin M (IgM)) or anti-hepatitis C virus (HCV)-test
19. Current drug or alcohol dependence
20. Blood donation (including donation of plasma and platelets) or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the patient
21. Participation in an interventional clinical trial during the last 2 months prior to individual enrolment of the patient
22. Patients who report a frequent occurrence of migraine attacks (i.e. at least once per month)
23. History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
24. Change in habits of physical activity within the last 2 months for at least 7 days (e.g. immobilisation due to bed rest, immobilisation of a leg or other big muscle groups)
25. Positive pregnancy test at screening examination
26. Pregnant or lactating women
27. Not willing to apply highly effective contraceptive methods [i.e. combined (estrogen and progestogen containing) hormonal contraception e.g. oral, intravaginal, transdermal and progestogen-only hormonal contraception e.g. oral, injectable, implantable as well as intrauterine device (IUD) and intrauterine hormone-releasing system (IUS) in combination with male condom; bilateral tubal occlusion, vasectomised partner or sexual abstinence]
28. Patients suspected or known not to follow instructions
29. Patients who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Impact of Ketosteril® on the generation of nitrogenous waste products | 10 days
  Serum urea
Impact of Ketosteril® on the generation of nitrogenous waste products | 10 days
  Urine urea
Impact of Ketosteril® on the generation of nitrogenous waste products | 10 days
  Nitrogen balance
Impact of Ketosteril® on the generation of nitrogenous waste products | 10 days
  Normalized protein catabolic rate (nPCR)
Protein metabolism | 10 days
  Serum total proteins
Protein metabolism | 10 days
  Albumin
Protein metabolism | 10 days
  Transthyretin
Protein metabolism | 10 days
  Transferrin
Markers of anabolic signaling | 10 days
  Serum Insulin-like growth factor (IGF)-I
Markers of anabolic signaling | 10 days
  Insulin like growth factor (IGF)-II
Markers of anabolic signaling | 10 days
  IGF-binding protein 3

SECONDARY OUTCOMES:
Renal function | 10 days
  Proteinuria
Renal function | 10 days
  Albuminuria
Renal function | 10 days
  Serum and urine creatinine
Renal function | 10 days
  Serum and urine urea
Renal function | 10 days
  Serum urea nitrogen (SUN)
Renal function | 10 days
  Urine nitrogen
Renal function | 10 days
  Glomerular filtration rate estimated from serum creatinine (eGFR)
Renal function | 10 days
  Albumin-creatinine ratio
Renal function | 10 days
  Urea clearance
Nutritional status | 10 days
  Body weight
Nutritional status | 10 days
  Body Mass Index (BMI)
Nutritional status | 10 days
  Body composition (via Bio Impedance Spectroscopy)
Nutritional status | 10 days
  SUN-to-creatinine ratio
Glucose metabolism | 10 days
  Fasting blood glucose
Lipid profile | 10 days
  Triglycerides
Lipid profile | 10 days
  Cholesterol
Lipid profile | 10 days
  High-density lipoprotein (HDL)/Low-density lipoprotein (LDL)-cholesterol
Mineral status | 10 days
  Sodium
Mineral status | 10 days
  Calcium
Mineral status | 10 days
  Potassium
Mineral status | 10 days
  Magnesium
Mineral status | 10 days
  Phosphate (serum and urine)
Mineral status | 10 days
  Alkaline phosphatase
Mineral status | 10 days
  Fibroblast growth factor (FGF)-23
Mineral status | 10 days
  25-hydroxycholecalciferol (serum)
Acid-base balance | 10 days
  Serum bicarbonate
Acid-base balance | 10 days
  Arterialized venous blood potential of hydrogen (pH)
Acid-base balance | 10 days
  Urine pH
Inflammation | 10 days
  Serum C-reactive protein (CRP)
Inflammation | 10 days
  Serum albumin/CRP ratio
Hematology | 10 days
  Hematocrit
Hematology | 10 days
  Hemoglobin
Hematology | 10 days
  Red blood cell (RBC) count
Hematology | 10 days
  White blood cell (WBC) count total
Hematology | 10 days
  WBC count differential (lymphocytes, basophils, monocytes, neutrophils, eosinophils)
Hematology | 10 days
  Platelet count
Hematology | 10 days
  Mean corpuscular hemoglobin (MCH)
Hematology | 10 days
  Mean corpuscular hemoglobin concentration (MCHC)
Hematology | 10 days
  Mean corpuscular volume (MCV)
Coagulation | 10 days
  Prothrombin time (Quick)
Coagulation | 10 days
  Activated partial thromboplastin time (APTT)
Coagulation | 10 days
  International normalized ratio (INR)
Serum chemistry | 10 days
  Glutamate oxaloacetate transaminase (GOT)/Aspartate aminotransferase (AST)
Serum chemistry | 10 days
  Glutamate-pyruvate transaminase (GPT)/Alanine transaminase (ALT)
Serum chemistry | 10 days
  Uric acid
Serum chemistry | 10 days
  Creatine kinase (CK)
Serum chemistry | 10 days
  Troponin T if CK is elevated
Serum chemistry | 10 days
  Chloride
Adverse Events | 52 days
  Adverse Events
Vital signs | 10 days
  Systolic and diastolic blood pressure
Vital signs | 10 days
  Pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: John F Stover, M.D., Study Chair — Fresenius Kabi
Locations (1):
- Thomayer Hospital Clinical - Pharmacology Unit (CPU), Prague, Czechia

IPD SHARING:
Plan to Share IPD: No